CLINICAL TRIAL: NCT01738529
Title: Characterization of Crohn's Disease at Confocal Laser Endomicroscopy and Related to Disease Activity
Brief Title: Characterization of Crohn's Disease at Confocal Laser Endomicroscopy (CLE) and Related to Disease Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, John Gasdal Karstensen, MD., Herlev Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-1-2012-089 sub 3
Record Dates: First submitted 2012-11-19; First posted 2012-11-30 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Crohn Disease
Keywords: confocal laser endomicroscopy; Crohn´disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLE ileocolonoscopy on Crohn patients (Active Comparator): Patients known with Crohn´s disease
  Interventions: Device: CLE ileocolonoscopy
- CLE ileocolonoscopy on control patients (Sham Comparator): CLE ileocolonoscopy on patients without known IBD
  Interventions: Device: CLE ileocolonoscopy

INTERVENTIONS:
Device: CLE ileocolonoscopy — The patients enrolled including the control group, will be investigated respectively, by conventional colonoscopy and CLE in both the terminal ileum as colon. The degree and extent of Crohn's disease are assessed by conventional ileocolonoscopy (SI), CLE (selected parameters) and histology biopsies. Then, the correlation between histology (gold standard), SI and CLE is calculated. An intra-and inter-observer study follows on CLE parameters, where 3 observers are blinded with respect to each other. The pathologist is blinded to conventional and CLE parameters. CLE results are stratified in order to identify which of the recorded CLE parameters that correlate best with the two other methods.
  Other Names: confocal laser endomiscoscopy ileocolonoscopy; confocal laser endomiscoscopy colonoscopy

SUMMARY:
A blinded prospective observation and methodology study with Confocal Laser Endomicroscopy (CLE) together with standard white light colonoscopy including inter- and intra-observation of patients with Crohn's disease.

DETAILED DESCRIPTION:
Introduction: Crohn's disease is a well-characterized disease, and treatment is carried out according to international guidelines. Despite this, the disease often show an individual, unpredictable course, and more than half of patients experience significant complications of the disease. Endoscopy is important for the assessment of disease dissemination and severity of Crohn's disease, which is complemented by biochemical and clinical indices, including CDAI or Simple Index (SI) (Harwey-Bradshaw), which is internationally recognized. By CDAI, there is shown a good correlation with the biochemical activity markers such as CRP, and serum albumin, and in practice the simplified version (SI). Is often used.

Knowledge about the use of CLE in Crohn's disease is very low. We will on the basis of parameters suggested in smaller studies and our personal CLE experience determine which parameters are useful for a precise estimation of the severity of Crohn's disease. Since the disease is most commonly seen in the terminal ileum, the parameters should apply to both the ileum and colon.

A group Crohn patients have long been in prolonged biochemical and conventional endoscopic remission, including patients treated with the biologic drug infliximab. These patients are also included in the study as a particularly interesting subgroup as CLE in a small study has suggested to contribute to the safe discontinuation of immunosuppressive therapy. The degree of healing of the mucous membrane including an intact barrier function is one of the most important prognostic factors for patients to develop a recurrence. Thus it will be of great clinical importance to clarify whether CLE can help to distinguish those patients who have an apparently normal endoscopy, yet unrealized discrete activity and defective barrier function from patients where there is no activity evaluated endoscopically and by CLE. Furthermore, a small number of patients will be included as a control group.

Hypothesis: CLE can characterize Crohn's disease and activity precisely in the ileum and colon compared with conventional ileocolonoscopy, including detecting slight degrees and wider dissemination of inflammation that would otherwise not be recognized.

Design: A blinded prospective observation and method study of patients with subsequent calculation of intra-and inter-observer variability.

Method: The patients enrolled including the control group, will be investigated respectively, by conventional colonoscopy and CLE in both the terminal ileum as colon. The degree and extent of Crohn's disease are assessed by conventional ileocolonoscopy (SI), CLE (selected parameters) and histology biopsies. Terminal ileum and each colonic segment (caecum, ascending colon, transversal colon, descending colon, colon sigmoid and rectum) are assessed as described above. Then, the correlation between histology (gold standard), SI and CLE is calculated. An intra-and inter-observer study follows on CLE parameters, where 3 observers are blinded with respect to each other. The pathologist is blinded to conventional and CLE parameters. CLE results are stratified in order to identify which of the recorded CLE parameters that correlate best with the two other methods, and thus are most suitable for the characterization and activity of Crohn's disease.

Statistical method: To calculate the CLE-finding in relation to respectively, SI and histology we use Spearman correlation analysis. At the inter-and intra-observer study used weighted Kappa.

Patient: A complete sample-size calculation has been made for the inter-and intra-observer study of the individual CLE parameters by 3 observers. For, if possible, to achieve a kappa value of 0.9 with a confidence interval of 0.05, there must be 122 observations. If we succeed in registering SI score, CLE parameters and taking tissue samples for pathology in all the above intestinal segments, there will be 7 observations for each patient who subsequently are assessed in relation to each of the parameters used in the study. If all ileocolonoscopy are completed and all CLE observations are possible to analyze just 18 patients need to be enrolled in the study. It is assumed, however, that there will only be 50% of the expected observations as some CLE observations will be unsatisfactory and some procedures will be interrupted. Thus, 36 patients shall be included in the study to achieve the desired strength, 10 of which are in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease and involvement of the ileum and / or colon
* Patients must be of legal age
* Shall be given written consent
* Both patients with the activity of their disease patients in remission on biological treatment including can be included
* The control group will consist of patients without known or suspected IBD

Exclusion Criteria:

* Increased p-creatinine
* Demonstrated allergy to fluorescein
* Pregnant woman
* Lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
CLE (CLE score) vs WL colonoscopy (SES-CD) | 1 year
  Findings in CLE are recorded regarding inflammation (crypt architecture, vessel architecture, barrier dysfunction and inflammatory cell invasion 1-3 points each) and compared with the findings of conventional colonoscopy ted Simple endoscopic score - Crohn´s disease (SES-CD), including observations for the control group
CLE (CLE-score) vs pathology score for inflammation | 1 year
  CLE (crypt architecture, vessel architecture, barrier dysfunction and inflammatory cell invasion 1-3 points each) and colonoscopy findings are compared with the pathological evaluation of the inflammation in the tissue samples (points from 1-3 by the severity).
CLE findings (CLE-score) and Intra-and inter-observer agreement | 1 year
  Intra-and inter-observer agreements between 3 operators at CLE findings are calculated by kappa statistics (crypt architecture, vessel architecture, barrier dysfunction and inflammatory cell invasion).

SECONDARY OUTCOMES:
Registering time of the procedure. | 1 year
  Registering time of the procedure.
Number of Adverse Events | 1 year
  Number of Adverse Events related to the procedure is registered

CONTACTS AND LOCATIONS:
Overall Officials: john g Karstensen, M.D., Principal Investigator — Department of Gastroenterology; peter vilmann, Prof., Study Chair — Department of Gastroenterology
Locations (1):
- Copenhagen University Hospital Herlev, Herlev, Denmark

REFERENCES:
- [Background] Kiesslich R, Duckworth CA, Moussata D, Gloeckner A, Lim LG, Goetz M, Pritchard DM, Galle PR, Neurath MF, Watson AJ. Local barrier dysfunction identified by confocal laser endomicroscopy predicts relapse in inflammatory bowel disease. Gut. 2012 Aug;61(8):1146-53. doi: 10.1136/gutjnl-2011-300695. Epub 2011 Nov 24. PMID 22115910
- [Background] Liu JJ, Wong K, Thiesen AL, Mah SJ, Dieleman LA, Claggett B, Saltzman JR, Fedorak RN. Increased epithelial gaps in the small intestines of patients with inflammatory bowel disease: density matters. Gastrointest Endosc. 2011 Jun;73(6):1174-80. doi: 10.1016/j.gie.2011.01.018. Epub 2011 Mar 11. PMID 21396639
- [Background] Li CQ, Xie XJ, Yu T, Gu XM, Zuo XL, Zhou CJ, Huang WQ, Chen H, Li YQ. Classification of inflammation activity in ulcerative colitis by confocal laser endomicroscopy. Am J Gastroenterol. 2010 Jun;105(6):1391-6. doi: 10.1038/ajg.2009.664. Epub 2009 Nov 24. PMID 19935787
- [Background] Vermeire S, Schreiber S, Sandborn WJ, Dubois C, Rutgeerts P. Correlation between the Crohn's disease activity and Harvey-Bradshaw indices in assessing Crohn's disease severity. Clin Gastroenterol Hepatol. 2010 Apr;8(4):357-63. doi: 10.1016/j.cgh.2010.01.001. Epub 2010 Jan 21. PMID 20096379
- [Background] Van Assche G, Dignass A, Reinisch W, van der Woude CJ, Sturm A, De Vos M, Guslandi M, Oldenburg B, Dotan I, Marteau P, Ardizzone A, Baumgart DC, D'Haens G, Gionchetti P, Portela F, Vucelic B, Soderholm J, Escher J, Koletzko S, Kolho KL, Lukas M, Mottet C, Tilg H, Vermeire S, Carbonnel F, Cole A, Novacek G, Reinshagen M, Tsianos E, Herrlinger K, Oldenburg B, Bouhnik Y, Kiesslich R, Stange E, Travis S, Lindsay J; European Crohn's and Colitis Organisation (ECCO). The second European evidence-based Consensus on the diagnosis and management of Crohn's disease: Special situations. J Crohns Colitis. 2010 Feb;4(1):63-101. doi: 10.1016/j.crohns.2009.09.009. Epub 2009 Dec 21. No abstract available. PMID 21122490
- [Derived] Karstensen JG, Saftoiu A, Brynskov J, Hendel J, Klausen P, Cartana T, Klausen TW, Riis LB, Vilmann P. Confocal laser endomicroscopy: a novel method for prediction of relapse in Crohn's disease. Endoscopy. 2016 Apr;48(4):364-72. doi: 10.1055/s-0034-1393314. Epub 2015 Nov 19. PMID 26583952